CLINICAL TRIAL: NCT04591626
Title: A Randomized, Double-Blind Trial Comparing the Effect of the Addition of Dulaglutide 1.5 mg Versus the Addition of Placebo to Titrated Basal Insulin on Glycemic Control in Chinese Patients With Type 2 Diabetes
Brief Title: A Study of Dulaglutide (LY2189265) in Chinese Participants With Type 2 Diabetes
Acronym: AWARD-CHN3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17731; H9X-MC-GBGO (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-10-16; First posted 2020-10-19 (Actual); Results first posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: T2DM; LY2189265
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 1.5 Milligrams (mg) Dulaglutide (Experimental): Participants received 1.5 mg Dulaglutide administered once weekly (QW) subcutaneously (SC) as add-on to titrated treat-to-target (TTT) dose of Insulin Glargine given SC, along with metformin and/or acarbose.
  Interventions: Drug: Dulaglutide; Drug: Insulin Glargine
- Placebo (Placebo Comparator): Participants received placebo administered QW SC as add-on to titrated TTT dose of insulin glargine given SC, along with metformin and/or acarbose.
  Interventions: Drug: Placebo; Drug: Insulin Glargine

INTERVENTIONS:
Drug: Dulaglutide — Administered SC
  Other Names: LY2189265
  Arms: 1.5 Milligrams (mg) Dulaglutide
Drug: Placebo — Administered SC
  Arms: Placebo
Drug: Insulin Glargine — Administered SC

SUMMARY:
The main purpose of this study is to evaluate the safety and efficacy of once weekly dulaglutide when added to insulin glargine, with metformin and/or acarbose in Chinese participants with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* have type 2 diabetes
* are men or nonpregnant women aged ≥18 years at screening
* have been treated with basal insulin glargine once daily and metformin and/or acarbose for at least 3 months prior to screening
* doses of once daily insulin glargine and OAMs must be stable during the 3-month period prior to screening. Insulin glargine dose is considered stable when all doses during this period are within the range defined by ±20% of the most commonly used insulin glargine dose during this same period. Doses of metformin and/or acarbose are considered stable when doses are unchanged during the same period, and the doses should be in the inclusive range of the half maximum to maximum approved daily dose per the locally-approved label
* have an HbA1c value ≥7.0% and ≤11.0% as assessed by the central laboratory at screening
* require further insulin glargine dose increase at baseline per the TTT algorithm based on the SMBG data (FBG ≥5.6mmol/L) collected during the prior week
* have stable weight (±5%) ≥3 months prior to screening
* have body mass index (BMI) between ≥19.0 and ≤35.0 kg/m2 at screening

Exclusion Criteria:

* have type 1 diabetes (T1D)
* have a history of ≥1 episode of ketoacidosis or hyperosmolar state/coma
* have a history of severe hypoglycemia and/or hypoglycemia unawareness within the 6 months prior to screening
* have had any of the following CV conditions within the 2 months prior to screening: acute myocardial infarction (MI), New York Heart Association (NYHA) Class III or Class IV heart failure, or cerebrovascular accident (stroke)
* have a known clinically significant gastric emptying abnormality (eg, severe diabetic gastroparesis or gastric outlet obstruction) or have undergone or plan to have a gastric bypass (bariatric) surgery or restrictive bariatric surgery (eg, Lap-Band®) during the course of the study, or chronically take drugs that directly affect gastrointestinal (GI) motility
* have a history of chronic pancreatitis or acute idiopathic pancreatitis, or were diagnosed with any type of acute pancreatitis within the 3 months prior to screening
* for participants on metformin or metformin and acarbose, have renal disease or renal dysfunction (eGFR [CKD-EPI] <45 mL/min/1.73 m2), as determined by the central laboratory; for participants on acarbose, have renal disease or renal dysfunction (eGFR [CKD-EPI] <25 mL/min/1.73 m2), as determined by the central laboratory
* have any self or family history of type 2A or type 2B multiple endocrine neoplasia (MEN 2A or 2B) syndrome in the absence of known C-cell hyperplasia (the only exception for this exclusion will be for participants whose family members with MEN 2A or 2B syndrome have a known RET mutation and the potential participant for the study is negative for the RET mutation)
* have any self or family history of medullary C-cell hyperplasia, focal hyperplasia, or carcinoma (including sporadic, familial, or part of MEN 2A or 2B syndrome)
* have serum calcitonin ≥20 pg/mL at screening, as determined by the central laboratory
* have any hematologic condition that may interfere with HbA1c measurement (eg, hemolytic anemias, sickle-cell disease)
* have been treated with any other antihyperglycemia regimen, other than basal insulin glargine once daily and metformin and/or acarbose, within the 3 months prior to screening or between screening and baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (27):
- China (27):
  - The Second People's Hospital of Hefei, Hefei, Anhui
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - First Affiliated Hospital of the Harbin Medical University, Harbin, Heilongjiang
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang Shi, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The First Hospital of Nanjing, Nanjing, Jiangsu
  - Nanjing Medical University - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - No. 2 Affiliated Hospital of Suzhou University, Suzhou, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - The Third Hospital of Nanchang, Nanchang, Jiangxi
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Dalian Municipal Central Hospital Affiliated of Dalian Medical University, Dalian, Liaoning
  - Jinan Central Hospital, Jinan, Shandong
  - Shanghai Putuo District Center Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Medical University, Xi’an, Shanxi
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The Affiliated Jiangyin Hospital of Southeast University Medical College, Wuxi, Wuxi Shi
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - Chongqing General Hospital, Chongqing, Yuzhong District
  - Zhejiang Hospital, Hangzhou, Zhejiang
  - Beijing Pinggu District Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1.5 Milligrams (mg) Dulaglutide | Placebo
Started | 144 | 147
Received At Least One Dose of Study Drug | 144 | 147
Completed | 134 | 142
Not Completed | 10 | 5
Not completed — Adverse Event | 4 | 0
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Death | 0 | 1
Not completed — Non-Compliance with Study Drug | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 1.5 mg Dulaglutide: Participants received 1.5 mg Dulaglutide administered QW SC as add-on to titrated TTT dose of insulin glargine given SC, along with metformin and/or acarbose.
- Total: Total of all reporting groups
Arm/Group | 1.5 mg Dulaglutide | Placebo | Total
Number analyzed (Participants) | 144 | 147 | 291
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.80 (9.33) | 58.30 (9.48) | 58.10 (9.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 57 | 109
  Male | 92 | 90 | 182
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 144 | 147 | 291
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 144 | 147 | 291
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 144 | 147 | 291
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time. Population: Participants with non-missing baseline value for HbA1c.
  Percentage of HbA1c
    number analyzed (Participants) | 136 | 145 | 281
    (all) | 8.60 (1.00) | 8.58 (0.97) | 8.59 (0.98)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time. Least Squares (LS) mean was determined by mixed model repeated measures (MMRM) model with Baseline + Oral Antihyperglycemic Medications (OAM) use + Treatment + Visit + Treatment*Visit (Type III sum of squares) as variables.
Time Frame: Baseline, Week 28
Population: All randomized participants with baseline and at least one post-baseline HbA1c data.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 1.5 mg Dulaglutide | Placebo
Number analyzed (Participants) | 133 | 142
Percentage of HbA1c | -2.03 (0.076) | -1.08 (0.073)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -0.95, 95% CI 2-sided [-1.14 to -0.77]

2. Secondary Outcome: Percentage of Participants Achieving HbA1c <7.0%
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time. Odds Ratio (OR) was determined using longitudinal logistic regression model with Baseline HbA1c value + OAM use + Treatment + Visit + Treatment*Visit as variables.
Time Frame: Week 28
Population: All randomized participants with baseline and at least one post-baseline HbA1c data.
Measure: Number; unit: Percentage of participants
Arm/Group | 1.5 mg Dulaglutide | Placebo
Number analyzed (Participants) | 133 | 142
Percentage of participants | 75.9 | 33.8
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 10.91, 95% CI 2-sided [5.35 to 22.28]

3. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight was reported here. LS mean was determined by MMRM model with Baseline + Baseline HbA1c strata (<8.5%, >=8.5%) + OAM use + Treatment + Visit + Treatment*Visit (Type III sum of squares) as variables.
Time Frame: Baseline, Week 28
Population: All randomized participants with baseline and at least one post-baseline body weight data.
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | 1.5 mg Dulaglutide | Placebo
Number analyzed (Participants) | 133 | 142
kilogram (kg) | -0.76 (0.224) | 0.42 (0.217)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -1.18, 95% CI 2-sided [-1.77 to -0.60]

4. Secondary Outcome: Change From Baseline in Fasting Serum Glucose (FSG)
Description: Change from baseline in FSG was reported here. LS mean was determined using MMRM model with Baseline + Baseline HbA1c strata (<8.5%, >=8.5%) + OAM use + Treatment + Visit + Treatment*Visit (Type III sum of squares) as variables.
Time Frame: Baseline, Week 28
Population: All randomized participants with baseline and at least one post-baseline fasting serum glucose data.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | 1.5 mg Dulaglutide | Placebo
Number analyzed (Participants) | 133 | 142
milligrams per deciliter (mg/dL) | -58.47 (2.339) | -43.64 (2.269)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -14.82, 95% CI 2-sided [-20.57 to -9.08]

5. Secondary Outcome: Percentage of Participants Achieving HbA1c <7.0% With no Weight Gain (<0.1 kg) and Without Documented Symptomatic Hypoglycemia (Blood Glucose <3.0 mmol/L)
Description: Percentage of Participants Achieving HbA1c <7.0% With no Weight Gain (<0.1 kg) and Without Documented Symptomatic Hypoglycemia (Blood Glucose <3.0 mmol/L) was reported here.
Time Frame: Week 28
Population: All randomized participants with HbA1c, hypoglycemia and body weight data.
Measure: Number; unit: Percentage of participants
Arm/Group | 1.5 mg Dulaglutide | Placebo
Number analyzed (Participants) | 139 | 147
Percentage of participants | 51.8 | 21.1
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.58, 95% CI 2-sided [2.64 to 7.95] — OR was determined using Logistic Regression model with Baseline HbA1c value + OAM use + Treatment as variables

6. Secondary Outcome: Percentage of Participants Achieving HbA1c <7.0% Without Documented Symptomatic Hypoglycemia (Blood Glucose <3.0 mmol/L)
Description: Percentage of Participants Achieving HbA1c <7.0% Without Documented Symptomatic Hypoglycemia (Blood Glucose <3.0 mmol/L) was reported here.
Time Frame: Week 28
Population: All randomized participants with HbA1c and hypoglycemia data.
Measure: Number; unit: Percentage of participants
Arm/Group | 1.5 mg Dulaglutide | Placebo
Number analyzed (Participants) | 139 | 147
Percentage of participants | 74.8 | 33.3
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 7.59, 95% CI 2-sided [4.27 to 13.48] — OR was determined using logistic regression model: Variable = Baseline HbA1c value + OAM use + Treatment as variables

7. Secondary Outcome: Percentage of Participants Achieving HbA1c <7.0% Without Weight Gain (<0.1 kg)
Description: Percentage of Participants Achieving HbA1c <7.0% Without Weight Gain (<0.1 kg) was reported here.
Time Frame: Week 28
Population: All randomized participants with HbA1c and body weight data.
Measure: Number; unit: Percentage of participants
Arm/Group | 1.5 mg Dulaglutide | Placebo
Number analyzed (Participants) | 139 | 147
Percentage of participants | 51.8 | 21.1
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.58, 95% CI 2-sided [2.64 to 7.95] — OR was determined using logistic regression model with Baseline HbA1c value + OAM use + Treatment as variables

8. Secondary Outcome: Change From Baseline in Blood Glucose From Daily Self-Monitored Blood Glucose (SMBG) Profile
Description: The SMBG data was collected at the following 7 time points: Pre morning meal BG, 2-hour postprandial measurement for morning meal BG, Pre midday meal BG, 2-hour postprandial measurement for midday meal BG, Pre evening meal BG, 2-hour postprandial measurement for evening meals BG, and Bedtime BG. LS mean was determined using MMRM model with Baseline + OAM (metformin and/or acarbose) usage + HbA1c Group at Baseline + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 28
Population: All randomized participants with baseline and at least one post-baseline blood glucose data from SMBG profile.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | 1.5 mg Dulaglutide | Placebo
Number analyzed (Participants) | 125 | 132
milligrams per deciliter (mg/dL) | -64.0 (2.42) | -37.7 (2.36)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -26.3, 95% CI 2-sided [-33.0 to -19.6]

9. Secondary Outcome: Change From Baseline in Daily Mean Insulin Glargine Doses
Description: LS mean was determined using MMRM model with Baseline + Baseline HbA1c strata (<8.5%, >=8.5%) + OAM use + Treatment + Visit + Treatment*Visit (Type III sum of squares) as variables.
Time Frame: Baseline, Week 28
Population: All randomized participants with a baseline and at least one post-baseline insulin glargine dose data.
Measure: Least Squares Mean (Standard Error); unit: International Units per day(IU/day)
Arm/Group | 1.5 mg Dulaglutide | Placebo
Number analyzed (Participants) | 133 | 143
International Units per day(IU/day) | 10.0 (1.045) | 14.0 (1.015)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Placebo; Test type: Superiority; p = 0.006, Mixed Models Analysis; LS Mean Difference = -4.0, 95% CI 2-sided [-6.86 to -1.14]

ADVERSE EVENTS:
Time Frame: Baseline Through End of Safety Follow-Up (Up To 32 Weeks)
Description: All randomized participants. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | 1.5 mg Dulaglutide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/144 | 1/147
Serious Adverse Events (participants affected / at risk) | 8/144 | 12/147
Other Adverse Events (participants affected / at risk) | 113/144 | 99/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.5 mg Dulaglutide (N=144) | Placebo (N=147)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Cataract nuclear (Eye disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Appendicolith (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 1.5 mg Dulaglutide (N=144) | Placebo (N=147)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 3 (3)
Ventricular extrasystoles (Cardiac disorders) | 2 (2) | 1 (1)
Thyroid mass (Endocrine disorders) | 2 (2) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 5 (6) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 11 (14) | 2 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 7 (9) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 19 (28) | 12 (25)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 8 (16) | 1 (1)
Flatulence (Gastrointestinal disorders) | 3 (4) | 0 (0)
Gastric dilatation (Gastrointestinal disorders) | 5 (6) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 15 (20) | 8 (8)
Toothache (Gastrointestinal disorders) | 5 (5) | 8 (11)
Vomiting (Gastrointestinal disorders) | 13 (14) | 2 (2)
Asthenia (General disorders) | 7 (12) | 1 (1)
Chest pain (General disorders) | 1 (1) | 2 (2)
Cyst (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 3 (3) | 4 (4)
Injection site reaction (General disorders) | 2 (4) | 0 (0)
Malaise (General disorders) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 2 (2)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Conjunctivitis (Infections and infestations) | 2 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Periodontitis (Infections and infestations) | 2 (2) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 11 (12) | 10 (15)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Vaginal infection (Infections and infestations) | 0/52 (0) | 2/57 (2)
Fractured coccyx (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Albumin urine present (Investigations) | 4 (4) | 2 (2)
Blood calcitonin increased (Investigations) | 0 (0) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 2 (2)
Blood pressure increased (Investigations) | 0 (0) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 2 (2)
High density lipoprotein decreased (Investigations) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 6 (6) | 2 (2)
Weight increased (Investigations) | 2 (3) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 32 (55) | 6 (6)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (5) | 11 (11)
Hyperlipidaemia (Metabolism and nutrition disorders) | 9 (9) | 7 (7)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Lipid metabolism disorder (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Osteoarthropathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/52 (0) | 1/57 (1)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 5 (7) | 6 (7)
Headache (Nervous system disorders) | 4 (4) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 2 (3)
Agitation (Psychiatric disorders) | 1 (2) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3)
Diabetic nephropathy (Renal and urinary disorders) | 20 (20) | 22 (22)
Microalbuminuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 2 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal cyst (Renal and urinary disorders) | 1 (1) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/92 (1) | 0/90 (0)
Cervical cyst (Reproductive system and breast disorders) | 0/52 (0) | 3/57 (3)
Fallopian tube obstruction (Reproductive system and breast disorders) | 0/52 (0) | 1/57 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 5 (5) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT04591626/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/26/NCT04591626/SAP_001.pdf